CLINICAL TRIAL: NCT03418935
Title: A Multicenter, Double-Blind, Placebo-Controlled, Randomized Trial of Efficacy and Safety of Remaxol®, a Solution for Intravenous Infusions Produced by STPF "POLYSAN" (Russia), in Patients With Mechanical Jaundice of Non-Malignant Origin
Brief Title: Remaxol® in Mechanical Jaundice of Non-malignant Origin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REM-OJ-III-16
Record Dates: First submitted 2018-01-19; First posted 2018-02-01 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Jaundice, Obstructive
Keywords: obstructive jaundice, non-malignant; mechanical jaundice, non-malignant; Methionine; Succinic acid
MeSH Terms: conditions — Jaundice, Obstructive | interventions — Remaxol; Succinic Acid; Methionine; Inosine; Niacinamide; Ringer's Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remaxol 400 ml (Experimental): Group I: treatment with Remaxol 400 ml IV + Ringer solution 400 ml IV for 7 days. Drug: Remaxol (succinate + methionine + inosine + nicotinamide)
  Interventions: Drug: Remaxol (succinate + methionine + inosine + nicotinamide); Drug: Ringer's Solution
- Remaxol 800 ml (Experimental): Group II: treatment with Remaxol 800 ml IV for 7 days. Drug: Remaxol (succinate + methionine + inosine + nicotinamide)
  Interventions: Drug: Remaxol (succinate + methionine + inosine + nicotinamide)
- Control (Placebo Comparator): Group III: Ringer's solution 800 ml IV for 7 days. Drug: Ringer's solution
  Interventions: Drug: Ringer's Solution

INTERVENTIONS:
Drug: Remaxol (succinate + methionine + inosine + nicotinamide) — Solution for intravenous infusions, containing succinate, methionine, inosine, and nicotinamide in 400 ml glass bottle
  Other Names: Remaxol®
  Arms: Remaxol 400 ml; Remaxol 800 ml
Drug: Ringer's Solution — Intravenous infusion, 400 or 800 ml
  Other Names: Placebo
  Arms: Control; Remaxol 400 ml

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Remaxol (succinate + methionine + inosine + nicotinamide; POLYSAN Ltd., Russia) infusions at dose 400 and 800 ml to treat mechanical jaundice of non-tumor cause during the first week after surgery.

DETAILED DESCRIPTION:
The study will be performed in in-hospital patients with obstructive jaundice cause by conditions other than tumor (predominantly by cholelithiasis; ICD-10 codes K80 and K83.1). The patients will be screened in the 15 days preceeding the appointed drainage surgery. The treatment will be started in the first 6 hours after the drainage surgery and continue for 7 days.

Following screening, patients who meet the inclusion criteria and have no criteria for exclusion will be randomly assigned into three study groups in the proportion of 1: 1: 1):

Group I: treatment with Remaxol 400 ml IV + Ringer solution 400 ml IV for 7 days.

Group II: treatment with Remaxol 800 ml IV for 7 days. Group III (control): Ringer solution 800 ml IV for 7 days.

Physical examination data, vital signs, biochemistry panel (including bilirubin, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, GGTP) will be assessed on days 1-8, on day 11 and day 14.

Diagnostic abdominal ultrasound will be performed before surgery and on days 3 and 8.

Neurophysiological test for the evaluation of the degree of encephalopathy will be performed before surgery, on days 3, 5, 8, and 14.

All patients will be followed up for 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of signed informed consent for participation in the study.
2. Men and women over the age of 18 (incl.).
3. Obstructive jaundice, verified by enlargement of intrahepatic bile ducts with proven non-tumor obstruction of extrahepatic bile ducts.
4. Duration of mechanical jaundice 15 days or less.
5. The level of total bilirubin in the blood from 5-fold to 20-fold exceeding normal.
6. Laboratory data corresponding to the following cutoff limits :

   * hemoglobin ≥90 g / l;
   * neutrophils ≥ 1.5x109 / l;
   * Platelets ≥ 75 x 109 / L;
   * AsAT and / or AlAT above 3 х normal but less than 20 х normal
   * Serum creatinine not exceeding 2 × normal,
   * Serum potassium within normal limits
7. Negative urine test for pregnancy in women of reproductive age.
8. Consent to use adequate methods of contraception or for complete abstinence from sexual activity for the period of the study.
9. Consent to abstain completely from alcohol intake during the study period.

Exclusion Criteria:

1. Tumor causing the obstruction of the bile ducts or the presence of any other malignancy at the time of randomization.
2. The need for another radical surgery within 2 weeks from the planned date of randomization.
3. Acute destructive pancreatitis, diffuse or diffuse peritonitis, sepsis.
4. Preexisting liver cirrhosis.
5. Exacerbation of the chronic peptic ulcer.
6. Ongoing bleeding.
7. Presence of clinically significant cardiovascular diseases: chronic cardiac insufficiency III-IV functional class by NYHA, uncontrolled arterial hypertension, acute stroke or acute myocardial infarction in the previous 3 months, unstable angina, uncontrolled arrhythmia and severe heart rhythm disturbances.
8. Any other decompensated disease.
9. Pregnancy or lactation.
10. Hypersensitivity to any component of the study drug / placebo and / or intolerance to any component of the study drug / placebo.
11. Regular admission of medications prohibited or not permitted by the study protocol within 4 weeks prior to enrollment.
12. Concomitant chronic systemic immune or hormonal therapy.
13. Gout.
14. Alcohol and/or drug dependence.
15. Active tuberculosis, HIV infection, syphilis, acute viral hepatitis.
16. Any other conditions / diseases that may interfere with the patient's compliance with the requirements of the Protocol.
17. Mental, physical and other reasons that do not allow the patient to comply with the requirements of the study protocol.
18. Any other significant (by judgement of the investigator) condition that prevents the patient from entering the study.
19. Participation in any clinical trial in the previous 3 months.
20. Staff of the research center and their family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Days to regression of jaundice | 14 days
  Time (days) from the date of drainage surgery to the reduction of the total bilirubin level down to 50 μmol / l, in experimental (Remaxol®) and control (Placebo) groups

SECONDARY OUTCOMES:
Disappearance of cytolysis (normal alanine aminotransferase and aspartate aminotransferase serum levels) on day 5 | 5 days
  Proportion of patients in study groups who reached normal serum levels of alanine aminotransferase and aspartate aminotransferase on day 5 from the start of treatment
Disappearance of cholestasis on day 5 | 5 days
  Proportion of patients in study groups who reached normal serum levels of alkaline phosphatase, GGTP, total bilirubin, and direct bilirubin on day 5 from the start of treatment
Disappearance of encephalopathy on day 5 | 5 days
  Proportion of patients in study groups who had normal brain functioning on day 5, as reflected by the neurophysiological test for the evaluation of the degree of encephalopathy
Serum bilirubin | 14 days
  Dynamics of total and direct bilirubin serum levels against baseline values and between visits in the study groups
Serum enzymes | 14 days
  Dynamics of serum alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, and GGTP against baseline values and between visits in the study groups
Liver function | 14 days
  State of liver protein synthesis function (as reflected by serum levels of total protein, albumin, fibrinogen) against baseline values and/or between visits
Kidney function | 14 days
  State of kidney function (serum creatinine) against baseline values and/or between visits
Proportion of patients with complications of jaundice | 14 days
  The number of patients in the study groups who developed complications in the postoperative period which were, according to the researcher's assessment, causally related to the obstructive jaundice (for example, purulent cholangitis, sepsis, kidney failure).

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail S. Bogomolov, MD, PhD, Study Director — St. Petersburg State Medical University n.a. I.P.Pavlov.
Locations (13):
- Russia (13):
  - Moscow 'City Clinical Hospital #24, Moscow
  - Moscow City Clinical Hospital #1 n.a.N.I.Pirogov, Moscow
  - Moscow City Clinical Hospital #29 n.a.N.A.Bauman, Moscow
  - Moscow City Clinical Hospital #67 n.a. L.A.Vorohobova, Moscow
  - Novosibirsk State Medical University, Novosibirsk
  - City Clinical Hospital of Emergency Care, Ryazan
  - North-West State Medical University named after I.I. Mechnikov, Saint Petersburg
  - State Budgetary Health Care Institution "City Hospital № 26", Saint Petersburg
  - Hospital for War Veterans, Saint Petersburg
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Saint-Petersburg I.I.Dzanelidze Research Institute of Emergency Medicine, Saint Petersburg
  - City Clinical Hospital #3 n.a.B.I.Alperovich, Tomsk
  - GBUZ YO 'Regional Clinical Hospital', Yaroslavl

IPD SHARING:
Plan to Share IPD: No